CLINICAL TRIAL: NCT05136937
Title: An Open-Label, Dose Escalation Study of the Safety and Tolerability of Oncolytic Virus Injection(RT-01) When Administered Via Intratumoral Injection in Patients With Advanced Solid Tumors
Brief Title: A Clinical Study of Intratumoral Administration of RT-01 in Patients With Advanced Solid Tumors
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Wuxi People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: LWY21076C1
Record Dates: First submitted 2021-11-01; First posted 2021-11-30 (Actual); Last update posted 2022-01-31 (Actual); Status verified 2022-01

CONDITIONS: Solid Tumor; Advanced Cancer
Keywords: RT-01; immunotherapy; intratumoral injection; oncolytic virus

STUDY DESIGN:
Intervention Model Description: Administered by intratumoral injection for 3 dose cohorts: 1×10^7 TCID50/mL, 1×10^8 TCID50/mL and 5×10^8 TCID50/mL
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Oncolytic virus injection(RT-01) for patients with advanced solid tumors (Experimental): Intratumoral administration of RT-01 as single agent for patients with advanced solid tumors.The injection dose of RT-01 was determined by the lesion size:
  1. mL for lesion length <1.5 cm;
  2. mL for lesion length between 1.5 cm and 2.5 cm;
  3. mL for lesion length between 2.5 cm and 5.0 cm;
  4. mL for lesion length between >5 cm
  Interventions: Biological: Oncolytic Virus Injection(RT-01)

INTERVENTIONS:
Biological: Oncolytic Virus Injection(RT-01) — Administered by intratumoral injection for 3 dose cohorts: 1×10^7 TCID50/mL, 1×10^8 TCID50/mL and 7×10^8 TCID50/mL

SUMMARY:
This is an open-label, dose escalation study of the safety and tolerability of oncolytic virus injection(RT-01) when administered via intratumoral injection in patients with advanced solid tumors. The purpose of this study is to assess the safety and tolerability of RT-01 and to determine the recommended phase 2 dose (RP2D) for further study. The study will also evaluate antitumor activity, objective response rate, pharmacokinetics and virus shedding of RT-01.

DETAILED DESCRIPTION:
This is an investigator initiated , open-label, study of RT-01 given via intratumoral (IT) injection as a single agent in participants with advanced solid tumors. The study is a single agent dose escalation which will use a 3+3 design to evaluate escalating doses of RT-01. Total enrollment will depend on the toxicities and/or activity observed, with approximately 7-18 evaluable participants enrolled.

The primary study objective is to determine the safety, tolerability, and maximum tolerated dose (MTD) of intratumoral administration of RT-01 as a single agent. Secondary objectives will assess efficacy overall response rate, as well as disease control rate, progression free survival, duration of response, and anti-tumor immune responses.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged ≥ 18 years;
* Subjects must have histologically- or cytologically-confirmed diagnosis of advanced solid tumor(s) and have progressed on or is not eligible for available standard therapy;
* Subjects have At least one measurable lesion according to Response Evaluation Criteria in Solid Tumors (RECIST 1.1) (non-nodal lesions with longest diameter ≥ 10 mm, or nodal lesions with short diameter ≥ 15 mm);
* ECOG score of 0 ~ 2;
* Adequate bone marrow, hepatic and renal and coagulation function;
* Women of childbearing age who have a negative pregnancy test within 7 days before treatment. Female patients of childbearing age, and male patients with partners of childbearing age must agree to use at least one medically recognized contraceptive method during study treatment and within at least 6 months after the last dose of investigational drug;
* Voluntarily participated in this study, signed the informed consent form, had good compliance, and cooperated with the follow-up.

Exclusion Criteria:

* Subjects with known brain metastasis and/or clinically history tumor brain of metastasis；
* Subjects who have received anti-tumor therapy such as chemotherapy, radiotherapy, biological therapy, endocrine therapy, targeted therapy, immunotherapy, etc within 4 weeks；
* Subjects who have participate in another interventional study while receiving study IP within 4 weeks；
* Subjects who have had major surgery ≤ 4 weeks of dosing；
* Patients in any condition requiring systemic treatment with corticosteroids (prednisone > 10 mg/day or equivalent of the similar drug) or other immunosuppressive agents within 14 days prior to investigational drug administration, but currently or previously treated with any of the following steroid regimens, were included:

  * Topical, ophthalmic, intra-articular, intranasal, or inhaled corticosteroids with minimal systemic absorption;
  * Prophylactic short-term (≤ 7 days) use of corticosteroids (e.g., allergy to contrast media) or for the treatment of non-autoimmune diseases (e.g., delayed hypersensitivity caused by contact allergens)
* Subjects received live vaccines within 7 days of initiation of study treatment；
* Subjects with adverse reactions caused by previous anti-tumor treatment not recovered to (CTCAE 5.0) grade 1 (except alopecia)；
* Subjects who have any active infection；
* Subjects with known positive history of human immunodeficiency virus (HIV) test or known acquired immunodeficiency syndrome (AIDS)；
* Subjects who have active hepatitis；
* Subjects who have serious cardiovascular system disorders history；
* Subjects with active autoimmune diseases or history of autoimmune diseases that may relapse；
* Subjects having any serious uncontrolled disease or in other conditions that would preclude them from receiving study treatment and are considered unsuitable for this study in the opinion of the investigator.
* Subjects in other conditions that are considered unsuitable for this study by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2021-11-01 (Actual); Primary Completion 2022-06-01 (Estimated); Study Completion 2023-06-01 (Estimated)

PRIMARY OUTCOMES:
Dose Limiting Toxicities (DLT) | Up to 28 days
  To define the maximum tolerated dose (MTD) of intratumoral administration of RT-01 injection in humans with malignant tumors.

SECONDARY OUTCOMES:
Safety and tolerability assessed by Adverse Events (AEs) | Up to 6 months
  An AE is any untoward medical occurrence in a subject administered an investigational product (IP), and which does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of IP whether or not considered related to the IP
Number of participants with laboratory value abnormalities and/or adverse events | Up to 6 months
  Number of participants with potentially clinically significant laboratory values
Number of participants with vital sign abnormalities and /or adverse event | Up to 6 months
  Number of participants with potentially clinically significant vital sign values
Safety assessed by 12- lead electrocardiograms (ECGs) adverse events | Up to 6 months
  12-lead ECGs will be read and assessed locally. Any clinically significant adverse changes on the ECG will be reported as Adverse Events
To evaluate the efficacy assessed per RECIST and iRECIST | Up to 2 years form first dose of RT-01
  Changes in tumor size and occurrence of metastases was assessed by the Response Evaluation Criteria in Solid Tumors (RECIST). Complete Response is disappearance of all target lesions. Partial Response is at least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum of diameters. Progressive Disease is at least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). And Stable Disease is neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum of diameters while on study.
Number of Participants With Response | at baseline, 2, 4, 7, 14, 28 days after injection
  Detection of increased systemic immune Response markers in peripheral blood mononuclear cells
Viral shedding of RT-01 in blood | Up to 6 months
  Viral DNA will be analyzed by quantitative polymerase chain reaction (qPCR).
Presence of neutralizing antibodies of antidrug antibodies (ADAs) development | Up to 6 months
  To evaluate the immunogenicity of RT-01 given as single agent post injection

CONTACTS AND LOCATIONS:
Locations (1):
- Wuxi People's Hospital, Wuxi, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No